CLINICAL TRIAL: NCT07307508
Title: Efficacy of Scalp Block in Managing Post Subarachnoid Hemorrhage Headache in Critically Ill Patients. A Single Centre Randomized Controlled Trial
Acronym: SAH-BLOCK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MRC-01-23-789; MRC-01-23-789 (Other Grant/Funding Number: Hamad Medical Corporation)
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage (aSAH); Headache Disorders
Keywords: Subarachnoid Hemorrhage Headache; Aneurysmal Subarachnoid Hemorrhage; Cerebral Aneurysm; SAH-associated headache; Scalp Block; Levobupivacaine; Opioid Consumption; Neurocritical Care
MeSH Terms: conditions — Subarachnoid Hemorrhage; Headache Disorders; Intracranial Aneurysm

STUDY DESIGN:
Intervention Model Description: The study involves a two-arm, randomized, parallel assignment. Recruited patients in the intervention group will receive a scalp block using 20 ml of 0.5% Levobupivacaine, while the control group will not receive any scalp block. The scalp block will be performed using an aseptic technique by a privileged anesthesiologist or intensivist after the endovascular coiling, while the patient is under general anesthesia, before extubation. All patients enrolled in the study will be blinded to the group randomization. However, the investigators will not be blinded to group assignments.
Who Masked: Participant
Masking Description: All patients enrolled in the study will be blinded to the group randomization. However, the investigators will not be blinded to group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Scalp Block with Levobupivacaine) (Experimental): Patients randomized to the intervention group will receive a scalp block using 20 ml of 0.5% Levobupivacaine after endovascular intervention and before extubation. In addition to conventional pain managment
  Interventions: Procedure: Levobupivacaine Scalp block
- Control arm (Active Comparator): Patients in the control group will receive no scalp block. Only conventional pain management will be given
  Interventions: Other: Conventional analgesic therapy

INTERVENTIONS:
Procedure: Levobupivacaine Scalp block — Scalp block will be administered using 20 ml of 0.5% Levobupivacaine In addition to conventional analgesic therapy. It will be performed using an aseptic technique by a privileged anesthesiologist or intensivist after the endovascular coiling, while the patient is under general anesthesia, before extubation. The scalp block will be administered using anatomical landmarks over the supraorbital and supratrochlear nerve, auriculotemporal nerve, zygomaticotemporal nerve, greater occipital nerve, and lesser occipital nerve.
  Arms: Intervention arm (Scalp Block with Levobupivacaine)
Other: Conventional analgesic therapy — The control group will recieve conventional therapy comprising regular intravenous paracetamol 1 gram every 6 hours intravenously plus fentanyl patient-controlled analgesia
  Arms: Control arm

SUMMARY:
Subarachnoid hemorrhage (SAH) is a devastating neurological disorder associated with significant mortality and morbidity rates, arising not just from the hemorrhage itself but also because of the catastrophic multisystem sequelae that can accompany the condition.

Rupture of an intracranial aneurysm accounts for up to 85% of instances of SAH, occurring in approximately 3 to 25 people per 100,000 annually in most populations. Treatment of aneurysmal SAH (aSAH) includes prevention of re-bleeding, evacuation of space-occupying hematomas, management of hydrocephalus, and prevention of secondary cerebral insult. Severe headache is the predominant characteristic symptom of aSAH, developing almost instantaneously at ictus in 50% of cases and continuing into the first days. Its severity has a variety of physiological and psychological effects on the patient. Scalp blocks have been suggested to alleviate this headache in case series. However, there is no strong evidence supporting this intervention. In this study, we aim to assess the impact of scalp blocks on headache reduction in patients undergoing endovascular treatment of an aneurysm (coiling or flow diversion) with aneurysmal subarachnoid bleeding.

DETAILED DESCRIPTION:
Despite its high prevalence, associated morbidity, and effects on the quality of life of aSAH-associated headache, epidemiological studies of its timing, severity, characteristics, and usual treatments are lacking. A prospective study in 2013 has shown that headache was the second-leading cause of 30-day hospital readmission after SAH. Long-term follow-up data indicate that headaches may persist after SAH for 2 to 9 years. Persistent headache leads to poor quality of life, increased therapy costs, delayed return to work, and increased incidence of depression.

Although there is evidence indicating that headaches related to subarachnoid hemorrhage (SAH) result in hospital readmissions and cause long-term suffering, there is a lack of data guiding the management of headaches in the critical care setting. Current national and international guidelines from the American Heart Association and the Neurocritical Care Society do not offer evidence-based recommendations for managing headaches. Furthermore, the exact mechanism of headache pain after subarachnoid hemorrhage remains elusive. Some researchers have postulated that this pain may be caused by hemolysis's inflammatory byproducts, resulting in meningeal irritation in the subarachnoid space. Additionally, central pain sensitization mediated by N-methyl-d-aspartate (NMDA) receptors may cause hyperalgesia after SAH. The lack of a definitive mechanism makes selecting Pharmacotherapeutics is a significant challenge. Innovative, opioid-sparing treatment strategies for managing SAH-associated headaches are warranted based on the need to monitor neurological examinations, avoid over-sedation, and alleviate discomfort in SAH patients with headaches. Opioids, often in escalating doses, remain the mainstay of therapy, in addition to other medications such as paracetamol, ketorolac, and dihydrocodeine. However, major limitations of this approach include depressed consciousness and respiratory drive, nausea, ileus, urinary retention, hypotension, and the high potential for tolerance and addiction. Headache management often remains suboptimal despite steady consumption of analgesics. Despite these obvious drawbacks, providers continue to rely on opioid therapy.

Review articles typically mention headaches after SAH without making specific Recommendations for managing the headache after the initial episode. However, a recent study evaluating Pterygopalatine Fossa Blockade (PPF) as a novel, narcotic-sparing treatment for headache in seven patients with SAH showed that the worst pain recorded in the 24 hours before the block was significantly higher than in the period four hours after the block (9.1 vs 3.1; p 0.0156), and in the period eight hours after the block (9.1 vs 2.8; = p 0.0313). The only complication was minor oozing from the needle insertion sites, which subsided completely with gauze pressure within 1 minute. In this study, we aim to assess the impact of scalp blocks in reducing headaches associated with aneurysmal subarachnoid hemorrhage in patients undergoing endovascular treatment of the aneurysm (coiling or flow diversion). To our knowledge, this will be the first randomized controlled trial to examine the role of scalp block in alleviating headaches associated with aSAH.

ELIGIBILITY:
Inclusion Criteria:

* All adults > 18 years who are admitted to the Surgical Intensive Care Unit (SICU) with a confirmed diagnosis of aneurysmal subarachnoid hemorrhage, undergoing endovascular treatment of the aneurysm (coiling/flow diversion).

Exclusion Criteria:

1. Patients with aSAH undergoing surgical craniotomy and aneurysmal clipping.
2. Non-aneurysmal subarachnoid or other intracranial hemorrhage forms (e.g., Intracerebral hemorrhage).
3. SICU admission Glasgow Coma Scale (GCS) of 13 or lower.
4. WFNS Score 4 / 5 or requiring mechanical ventilation for more than 24 hrs.
5. Patients with known allergy to local anesthetics.
6. Admission to ICU > 7 days after hemorrhage.
7. Patients with a documented bleeding disorder.
8. Patients with a history of chronic headache disorder or migraine.
9. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Total opioid consumption in the first 24 hours after administration of scalp block. | 24 hours after intervention
  Total opioid dose administered within the first 24 hours following the scalp block + Standard care (intervention arm) Vs standard care alone (control arm). To calculate a uniform metric to quantify the daily total opioid dose per patient per day, the recorded amounts of the various opioid agents will be converted to their intravenous morphine equivalent by using standard conversion factors. The total resultant dosage will be calculated as the sum of all converted doses for each patient for each day in the study interval and presented as a morphine-equivalent dose. The maximum and median daily opioid dosage will be determined by examining these aggregated daily.

SECONDARY OUTCOMES:
Median numeric rating scores (NRS) pain scores in the first 24 hours after the administration of scalp block. | 24 hours after intervention
  Numeric Rating scores (NRS) is a tool to assess the severity of pain/headaches from zero to ten, where zero is no pain, and 10 is the worst pain possible. The patient-controlled analgesia (PCA) device is a device used to administer set doses of opioids with a safety lockout to prevent overdosing. However, the device is capable of registering the number of demands made by the patients even if no dose is delivered (i.e. demand made within lockout time). The recorded demand will be used as a surrogate for pain intensity

CONTACTS AND LOCATIONS:
Overall Officials: Sohel Mohamed Ahmed, Consultant, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to institutional policies at Hamad Medical Corporation and local regulatory restrictions. Only final results will be reported in publications and presentations.